CLINICAL TRIAL: NCT05864612
Title: Developing Interoperable Tools for Anxiety and Depression Screening in Epilepsy
Brief Title: Tools for Anxiety and Depression Screening in Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00086172; R03TR004251 (NIH)
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2024-09

CONDITIONS: Epilepsy
Keywords: anxiety; depression; screening tools
MeSH Terms: conditions — Epilepsy; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The four instrument delivery methods to be used in this pragmatic trial represent distinct prompts & cues for screening instrument completion. Examining these multiple instrument delivery methods will generate outputs that will support flexibility in instrument delivery modalities across multiple sites in future multicenter studies in this area. These 4 distinct delivery methods are used to deliver identical standard care validated anxiety and depression screening instruments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Text Message (Active Comparator): Subjects in this arm will be asked to complete standard care screening questionnaires on anxiety and depression, delivered by Twilio text message.
  Interventions: Behavioral: Screening Questionnaires
- Customized Email Prompt (Active Comparator): Subjects in this arm will be asked to complete standard care screening questionnaires on anxiety and depression, delivered by an email with a REDCap email survey link.
  Interventions: Behavioral: Screening Questionnaires
- Generic Electronic Health Record (EHR) portal email (Active Comparator): Subjects in this arm will be prompted with customized EHR portal message after login to EHR portal.
  Interventions: Behavioral: Screening Questionnaires
- EHR Portal with No Message (Active Comparator): Subjects in this arm will not receive a reminder, but previsit questionnaires associated with a visit will be in their EHR portal.
  Interventions: Behavioral: Screening Questionnaires

INTERVENTIONS:
Behavioral: Screening Questionnaires — Standard care screening questionnaires on anxiety and depression

SUMMARY:
A randomized trial to compare patient-completion success of REDCap and Electronic Health Record (EHR)-based anxiety & depression instrument delivery methods. Study hypothesis is that the screening completion proportion will vary across the 4 modalities tested.

DETAILED DESCRIPTION:
In this randomized study of four modalities, we will compare Twilio text message delivery via REDCap versus (vs.) REDCap email survey links vs. EHR portal questionnaires with reminder message vs. current standard delivery EHR portal questionnaires without reminder. Screening instruments will be delivered by randomized method 7 days prior to scheduled clinic visit and outcomes occur by the time of the scheduled clinic visit. The study setting is the Wake Forest Comprehensive Epilepsy Center, with 2 clinic sites where adult patients are served (Atrium Health Wake Forest Baptist main campus, Atrium Health High Point Medical Center). EHR portal questionnaires without reminder is the current standard care screener delivery method. An exploratory supplement randomizing individuals to text message versus email survey link was later added.

ELIGIBILITY:
Inclusion Criteria:

* Visit scheduled 7 days in advance at an adult-focused epilepsy clinic at the study site

Exclusion Criteria:

* No exclusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi M. Munger Clary, MD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and results published by primary study team, de-identified, archived data will be stored for potential use if requested by other qualified researchers including those outside of the study.
Supporting Information: Study Protocol, ICF
Time Frame: After the study is completed and results published, de-identified, archived data will be available upon request.

RESULTS

PARTICIPANT FLOW:
Groups:
- Electronic Health Record (EHR) Portal With No Message: Subjects in this arm will not receive a reminder, but previsit questionnaires associated with a visit will be in their EHR portal.
  Screening Questionnaires: Standard care screening questionnaires on anxiety and depression
Period: Overall Study
Arm/Group | Text Message | Customized Email Prompt | Generic Electronic Health Record (EHR) Portal Email | Electronic Health Record (EHR) Portal With No Message
Started | 221 | 221 | 219 | 219
Completed | 221 | 221 | 219 | 219
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text Message | Customized Email Prompt | Generic Electronic Health Record (EHR) Portal Email | EHR Portal With No Message | Total
Number analyzed (Participants) | 221 | 221 | 219 | 219 | 880
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (16.9) | 42.3 (16.6) | 45.3 (18.1) | 41.2 (17.1) | 42.7 (17.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  male | 93 | 103 | 93 | 100 | 389
  female | 128 | 116 | 126 | 118 | 488
  unknown | 0 | 2 | 0 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 12 | 11 | 16 | 46
  Not Hispanic or Latino | 213 | 206 | 205 | 200 | 824
  Unknown or Not Reported | 1 | 3 | 3 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 2
  Asian | 2 | 3 | 1 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 38 | 49 | 47 | 38 | 172
  White | 173 | 155 | 157 | 158 | 643
  More than one race | 8 | 14 | 12 | 20 | 54
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Completing Screening Instruments
Description: Percentage of subjects completing screening instruments by each of the 4 methods prior to clinic visit will be used to compare the effect of the different methods on patient self-completion, and to estimate completion rates by different methods for use in future screening implementation trials.
Time Frame: Week 1
Measure: Number; unit: Percentage who completed
Arm/Group | Text Message | Customized Email Prompt | Generic Electronic Health Record (EHR) Portal Email | EHR Portal With No Message
Number analyzed (Participants) | 221 | 221 | 219 | 219
Percentage who completed | 0 | 14 | 19 | 12

2. Secondary Outcome: Research Team Time-sending Instruments
Description: Time in minutes will be recorded
Time Frame: Baseline Day 0
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Text Message | Customized Email Prompt | Generic Electronic Health Record (EHR) Portal Email | EHR Portal With No Message
Number analyzed (Participants) | 221 | 221 | 219 | 219
minutes | 3.0 (1.6) | 4.5 (1.8) | 1.7 (1.2) | 0.6 (0.6)

3. Secondary Outcome: Research Team Time-instrument Data Entry
Description: Time in minutes will be recorded
Time Frame: Week 1
Population: no responses received in Text Message Arm due to technical error in text delivery occurring outside of REDCap text sending interface
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Text Message | Customized Email Prompt | Generic Electronic Health Record (EHR) Portal Email | EHR Portal With No Message
Number analyzed (Participants) | 0 | 29 | 43 | 27
minutes |  | 2.5 (2.0) | 1.8 (2.0) | 1.7 (2.4)

4. Secondary Outcome: Participant Time From Instrument Delivery to Completion
Description: Time in minutes will be recorded
Time Frame: Week 1
Population: no responses received due to technical error in text delivery occurring outside of REDCap text sending interface - number of participants with instrument responses received - number of participants with instrument responses received - number of participants with instrument responses received
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Text Message | Customized Email Prompt | Generic Electronic Health Record (EHR) Portal Email | EHR Portal With No Message
Number analyzed (Participants) | 0 | 32 | 42 | 27
minutes |  | 4.6 (2.4) | 3.1 (2.6) | 2.2 (2.1)

5. Secondary Outcome: Percent Accuracy of Kit Application Programming Interface (API)
Description: Among participants who completed anxiety and depression screening instruments by one of the two EHR methods, this measure evaluates the % of instrument scores collected via Kit API that were identical to the original EHR source completion.
Time Frame: Week 1
Population: The analysis population for this outcome measure (accuracy of Kit API) is only participants randomized to one of the two EHR portal arms who also completed the pre-visit questionnaires and thus had questionnaires completed in the electronic health record available for testing Kit API data collection accuracy, as this tool is designed to collect data directly from the health record into REDCap.
Measure: Mean (Full Range); unit: percent scores identical to EHR source
Arm/Group | Text Message | Customized Email Prompt | Generic Electronic Health Record (EHR) Portal Email | EHR Portal With No Message
Number analyzed (Participants) | 0 | 0 | 43 | 27
percent scores identical to EHR source |  |  | 100 [100 to 100] | 100 [100 to 100]

6. Other Pre Specified Outcome: Clinic Visit Attendance:Visit Completed
Description: Number of visits completed out of number scheduled
Time Frame: Week 1
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Clinic Visit Attendance:Visit Canceled
Description: Number of visits completed out of number scheduled
Time Frame: Week 1
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Clinic Visit Attendance: No-show
Description: Number of no-show visits out of number scheduled
Time Frame: Week 1
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Time For Data Entry
Description: Time collected in minutes
Time Frame: Week 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Week 12
Arm/Group | Text Message | Customized Email Prompt | Generic Electronic Health Record (EHR) Portal Email | EHR Portal With No Message
All-Cause Mortality (participants affected / at risk) | 0/221 | 0/221 | 0/219 | 0/219
Serious Adverse Events (participants affected / at risk) | 0/221 | 0/221 | 0/219 | 0/219
Other Adverse Events (participants affected / at risk) | 0/221 | 0/221 | 0/219 | 0/219

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT05864612/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT05864612/ICF_001.pdf